CLINICAL TRIAL: NCT06369129
Title: Assessment of Accuracy and Orbital Volume Using Patient Specific Titanium Implant Vs Patient Specific Zirconia Implant for Orbital Floor Reconstruction in Blowout Fractures A Randomized Clinical Trial: Comparative Study
Brief Title: Accuracy& Orbital Volume Using Patient Specific Titanium Implant Vs Zirconia for Orbital Floor Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ola Alaa El-Din Abd El-Monem Mohamed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2024-06-16
Record Dates: First submitted 2024-04-06; First posted 2024-04-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Blow-Out Fractures; Orbital Fractures; Orbital Floor Fracture; Orbital Trauma
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial.
  * Parallel group study.
  * A trial will be carried out in hospital of Oral and Maxillofacial surgery department - Faculty of Oral and Dental Medicine - Cairo University .
  * Equal randomization : participants with equal probabilities for intervention.
  * Positive controlled : Both groups receiving treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orbital floor reconstruction with Patient Specific Zirconia Implant (Experimental): Orbital floor reconstruction with Patient Specific Zirconia Implant will be done
  Interventions: Procedure: Orbital floor reconstruction with Patient Specific Zirconia Implant
- Orbital floor reconstruction with Patient Specific Titanium Implant (Active Comparator): Orbital floor reconstruction with Patient Specific Titanium Implant will be done.
  Interventions: Procedure: Orbital floor reconstruction with Patient Specific Titanium Implant

INTERVENTIONS:
Procedure: Orbital floor reconstruction with Patient Specific Zirconia Implant — Orbital floor reconstruction with Patient Specific Zirconia Implant will be done
  Arms: Orbital floor reconstruction with Patient Specific Zirconia Implant
Procedure: Orbital floor reconstruction with Patient Specific Titanium Implant — Orbital floor reconstruction with Patient Specific Titanium Implant will be done
  Arms: Orbital floor reconstruction with Patient Specific Titanium Implant

SUMMARY:
Comparative study used to assess if the patient specific zirconia implant will provide better accuracy, intraoperative adaptability, precise orbital volume and soft tissue reaction with more cost effectiveness than the patient specific titanium implants in orbital floor reconstruction after blow out fractures .

DETAILED DESCRIPTION:
Patients of both groups will be subjected to:

1. Case history including personal data, medical, surgical history and family history.
2. A full examination of the cranial and maxillofacial skeleton and soft tissue .
3. Evaluation of Visual Functions
4. Ophthalmologic consultation and clearance
5. Radiographic examination: CT scan
6. All DICOM data will be imported to the surgical planning software.

Virtual planning:

1. A midsagittal plane will be constructed then the normal orbit will be mirrored to the affected side.
2. The mirrored orbital floor will be meshed with 1.6 mm holes then its peripheries will be extended downwards by 3 mm and meshed also in order to accommodate the fixation.
3. The designed part will be subtracted then exported in Stereolithography (STL) format to be fabricated .

   The surgery will be done under General anesthesia and undertaken within 14 days to prevent fibrosis. Can be delayed 24-72 hours to allow the edema to subside before undertaking surgery.

   Intervention Group: -

   • The STL file will be milled from zirconium and then will be ready for sterilization and intraoperative fixation

   - A transconjunctival incision will be done to allow for good exposure that optimizes visualization of the orbital floor during the repair and insertion and fixation of the patient specific zirconia implant.

   Control Group: -

   • The STL file be milled from grade 4 titanium and then will be ready for sterilization and intraoperative fixation with the same surgical steps.

   Follow up:

   All patients will be examined clinically and radiographically, during postoperative 1st and 2nd week .

   Only one postoperative CT scan will be done after 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with blow out fracture isolated and / or combined with other fracture.
* Age group: from 18 to 60 years old
* No sex predilection
* Patients with no contraindications to surgical intervention.
* Patients willing for the surgical procedure and follow-up, with an informed consent.

Exclusion Criteria :

* Medically compromised patients.
* Patients with history of previous orbital reconstruction surgery.
* Uncooperative patients.
* Patients with systemic contraindication to general anesthesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Orbital Volume | immediately post operative
  will be measured with CT scan in mm3

SECONDARY OUTCOMES:
Accuracy of the patient specific implant in the orbital floor reconstruction | immediately post operative
  will be measured with CT scan with superimposition of the preoperative CT scan and the mirrored image and the post operative CT scan . The difference will be measured by mm
Cost effectiveness | through study completion, an average of 1 year
  will compare between the prices of the patient specific implants the titanium and the zirconia and financial record will be kept with that in United states dollar . By the end of the study and comparison will be done to check which one was more cost effective
Patient satisfaction | through study completion, an average of 1 year
  will be assessed by a Questionnaire using Visual analogue scale , highest score will be more satisficed .The score is minimum 1 and maximum 10.

CONTACTS AND LOCATIONS:
Overall Officials: OLA A. ELMORSY, PHD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No